CLINICAL TRIAL: NCT04594928
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Efficacy of GLPG3667 in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Study Evaluating the Effects of GLPG3667 Given as an Oral Treatment for 4 Weeks in Adults With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GLPG3667-CL-112; 2020-001427-14 (EudraCT Number)
Record Dates: First submitted 2020-10-05; First posted 2020-10-20 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GLPG3667 Dose A (Experimental): Daily doses of GLPG3667 for 4 weeks.
  Interventions: Drug: GLPG3667
- GLPG3667 Dose B (Experimental): Daily doses of GLPG3667 for 4 weeks.
  Interventions: Drug: GLPG3667
- Placebo (Placebo Comparator): Placebo to match will be administered as capsules for daily oral use.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG3667 — GLPG3667 capsules
  Arms: GLPG3667 Dose A; GLPG3667 Dose B
Drug: Placebo — Matching placebo capsules
  Arms: Placebo

SUMMARY:
The purpose of this research study is to assess the safety, tolerability, efficacy, pharmacokinetics and pharmacodynamics of GLPG3667 in multiple daily oral doses in subjects with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be male or female between 18-64 years of age (extremes included), on the date of signing the informed consent form (ICF).
* Subject must be diagnosed (for at least 6 months before screening) of moderate to severe intensity plaque psoriasis. Subject's plaque psoriasis must be stable, defined as no flare during the month before the screening visit and no change of the severity between the screening visit and baseline visit.
* At screening and at baseline (Day 1, predose), PASI >=12 (moderate to severe) and plaque-type psoriasis covering at least 10% of total body surface area (BSA).
* At screening a Physician's Global Assessment (PGA ) score of 3 ("moderate") or 4 ("severe").
* Subject must be considered by dermatologist investigator to be a candidate for systemic therapy of plaque psoriasis (either naïve or history of previous systemic treatment).

This list only contains the key inclusion criteria.

Exclusion Criteria:

* Subject has a known hypersensitivity to investigational product (IP) ingredients or history of a significant allergic reaction to IP ingredients as determined by the investigator.
* Subjects with psoriasis other than plaque type or complicated psoriasis such as guttate, erythrodermic, exfoliative, inverse, pustular, palmo plantar, infected, or ulcerated psoriasis.
* Subject has evidence of skin conditions other than psoriasis (e.g. eczema) at the time of screening or baseline visit that would interfere with the evaluation of psoriasis.
* Subject is unable to discontinue prohibited therapies for the treatment of plaque psoriasis and/or cannot discontinue phototherapy (ultraviolet B (UVB) or psoralen and ultraviolet A (PUVA)) before the start of the study up to the end of the study.
* Subjects with current or a known or suspected history of immunosuppressive condition, history of invasive opportunistic infections (e.g. human immunodeficiency virus (HIV) infection, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis, or organ or bone marrow transplantation).
* Subjects having an active clinically significant infection or any infection requiring oral or systemic therapy within 2 weeks prior screening or subjects currently on any chronic oral or systemic antiinfective therapy for chronic infection.
* Subject testing positive for severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) infection as detected at screening based on real time polymerase chain reaction (RT-PCR) or at baseline based on Immunoglobulin M (IgM) immunoassay, or subjects who have been in contact with SARS-CoV-2 infected individuals in the two weeks prior to first dosing of IP. Subjects presenting any signs or symptoms of SARS-Cov-2 infection as detected at screening or baseline following careful physical examination (e.g. cough, fever, headaches, fatigue, dyspnea, myalgia, anosmia, dysgeusia, anorexia, sore throat, etc.). In addition, any other locally applicable standard diagnostic criteria may also apply to diagnose SARS-CoV-2 infection.
* Subjects with evidence of active or latent infection with Mycobacterium tuberculosis (TB) as defined by:

  1. Positive QuantiFERON-TB Gold test result, AND/OR
  2. Chest radiograph (posterior anterior view) taken within 12 weeks prior to screening, read by a qualified radiologist or pulmonologist, with evidence of current active TB or old inactive TB.
* Subjects with a history of TB who have successful treatment documentation are eligible for the study.

This list only contains the key exclusion criteria.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse events (SAEs), and TEAEs leading to treatment discontinuation in subjects with moderate to severe plaque psoriasis. | From screening through study completion, an average of 3 months
  To evaluate the safety and tolerability of GLPG3667 compared to placebo in subjects with moderate to severe plaque psoriasis.
Psoriasis Area and Severity Index (PASI) % change | At week 4
  To evaluate signs of clinical efficacy of GLPG3667 compared to placebo in subjects with moderate to severe plaque psoriasis.

SECONDARY OUTCOMES:
Observed GLPG3667 plasma trough concentrations (Ctrough). | Between Day 1 pre-dose and Day 30
  To characterize the pharmacokinetics (PK) of GLPG3667 in subjects with moderate to severe plaque psoriasis.
Change from baseline in interleukin 17 [IL-17] levels between treatment groups and time points. | Between Day 1 pre-dose and Day 60
  To evaluate blood pharmacodynamics (PD) markers in response to administration of GLPG3667 in subjects with moderate to severe plaque psoriasis.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Timmis, MD, Study Director — Galapagos NV
Locations (7):
- MC Comac Medical Ltd., Sofia, Bulgaria
- Poland (5):
  - Early Clinical Trials Unit University Clinical Centre, Gdansk
  - Barbara Rewerska Diamond Clinic Specjalistyczne Poradnie Lekarskie, Krakow
  - Centrum Medyczne All-Med, Lodz
  - Reumed Sp. z o. o., Lublin
  - WIP Warsaw IBD Point, Warsaw
- Summit Clinical Research, s.r.o., Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No